CLINICAL TRIAL: NCT06690606
Title: EOCRCPred: an AI Model for Predicting Overall Survival in Early-Onset Stage I-III Colorectal Cancer Patients Post-Radical Resection-A SEER Database and Dual-Center Chinese Medical Institutions Study
Brief Title: EOCRCPred: an AI Model to Predict Survival in EOCRC Patients After Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wanli Deng, MD, Principal Investigator, Shanghai University of Traditional Chinese Medicine
Other Study IDs: PTEC-A-2024-61 (S); 2021tszk01 (Other Grant/Funding Number: Health System of PuTuo District in Shanghai); 2023-BSH-02 (Other Grant/Funding Number: Putuo District Central Hospital)
Record Dates: First submitted 2024-11-12; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer
Keywords: AI model; prediction; Early-Onset Colorectal Cancer (EOCRC); postoperative survival; surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- external validation cohort: The external validation cohort was composed of primary EOCRC patients who underwent radical resection at Putuo Hospital and Yueyang Hospital, both affiliated with Shanghai University of Traditional Chinese Medicine. The cohort includes patients diagnosed between January 2014 and June 2024.
  Inclusion criteria: Patients with pathologically confirmed primary EOCRC, aged under 50 years, and who received radical surgery (stages I-III according to the AJCC 7th edition).
  Exclusion criteria: Patients with multiple primary cancers, survival time under 1 month, or missing critical data.

SUMMARY:
The goal of this observational study is to develop a predictive model for overall survival in patients under the age of 50 who have undergone surgery for early-onset colorectal cancer (EOCRC). The main question it aims to answer is:

Can machine learning models accurately predict the long-term survival of EOCRC patients after surgical treatment?

Participants who have already undergone surgery for EOCRC as part of their regular medical care will have their clinical data analyzed, with survival outcomes tracked through follow-up assessments. An online survival calculator will also be developed to aid clinicians and patients in predicting personalized survival outcomes.

DETAILED DESCRIPTION:
To avoid duplicating information that will be entered or uploaded elsewhere in the record, here is a concise summary of the key components of the study:

* Study Title**: *EOCRCPred: An AI Model to Predict Survival in Early-onset Colorectal Cancer Patients After Surgery*
* Introduction**:

This study addresses the increasing incidence and mortality of early-onset colorectal cancer (EOCRC) in patients under 50. EOCRC exhibits distinct clinical and pathological features compared to late-onset CRC, including higher recurrence rates and advanced disease stages at diagnosis. Current predictive models for postoperative outcomes in EOCRC are limited, highlighting the need for specialized tools to guide treatment decisions.

* Objectives**:

  1. Develop AI models for predicting overall survival (OS) in postoperative M0 EOCRC patients.
  2. Propose a new survival risk stratification system.
  3. Deploy an online survival calculator to assist clinical decision-making.
* Methods**:

  * **Data Source**: SEER database (2010-2019) for training/testing; two Chinese hospitals for external validation (2014-2024).
  * **Inclusion Criteria**: Pathologically confirmed primary EOCRC, radical surgery (stage I-III), and complete follow-up.
  * **Models**: Six predictive models, including CoxPH, RSF, S-SVM, XGBSE, GBSA, and DeepSurv.
  * **Evaluation Metrics**: Discrimination (C-index, time-dependent AUC), calibration (Brier score, calibration curves), and clinical utility (Decision Curve Analysis).
* Statistical Analysis**:

Comparisons were made using t-tests, Mann-Whitney U tests, and chi-square tests, with P < 0.05 indicating significance.

**Risk Stratification**: Risk groups were classified based on RSF-derived scores (low, intermediate, high), and survival differences were assessed via Kaplan-Meier curves and log-rank tests.

This streamlined summary covers the primary goals, methodology, and analysis without repeating specifics that will be detailed in other sections of the record.

ELIGIBILITY:
Inclusion Criteria:

* Primary EOCRC confirmed by pathological histological examination (ICD-10 codes: C18.0, C18.2-18.9, C19.9, C20.9)
* Radical surgery performed (Specific Surgery Codes 30-70, including partial/subtotal colectomy, hemicolectomy, right/left colectomy, and total colectomy, as well as partial or total removal of other organs and regional lymph nodes)
* Stage I-III disease according to the 7th AJCC-TNM system

Exclusion Criteria:

* Patients with multiple primary cancers or other malignancies
* Survival time of less than 1 month, or absence of postoperative follow-up information
* Incomplete critical clinical feature information

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive patients with early-onset, Stage I-III colorectal cancer who underwent radical resection at Putuo Hospital and Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, both affiliated with Shanghai University of Traditional Chinese Medicine, were retrospectively collected between January 2014 and June 2024.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-11-12 (Estimated); Primary Completion 2025-05-11 (Estimated); Study Completion 2025-05-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of Clinical Characteristics and Survival Status of Subjects Using the CRF Scale | 2024.11
  Age, Gender, Race, Primary Site, Tumor Diameter, Differentiation Degree, Histology, TNM Stage, CEA, Surgery Type, Number of Resected Lymph Nodes, Tumor Deposits, Neural Invasion, Radiation Sequence, Chemotherapy Sequence, Systemic Therapy Sequence, Marital Status, Household Income, Survival Status, Postoperative Survival Time.

CONTACTS AND LOCATIONS:
Overall Officials: Wanli Deng, Principal Investigator — Putuo Hospital, Shanghai University of Traditional Chinese Medicine
Locations (2):
- China (2):
  - Putuo Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share Individual Participant Data (IPD) has not been finalized due to several considerations. We are evaluating factors such as privacy and confidentiality risks, even with anonymization, as well as the ethical and legal implications of data sharing. Additionally, we must assess whether participants' consent allows for broader data sharing beyond the initial study purpose. These factors are under review, and a final decision will be made with careful consideration of participant protection and compliance with regulatory requirements.